CLINICAL TRIAL: NCT01504581
Title: A Randomized, Double-Blind, Placebo- And Active-Controlled Study Of The Pharmacokinetics, Pharmacodynamics And Safety Of Single Ascending Doses Of HM10660A (LAPS-INTERFERON ALPHA-2B) In Healthy Male Subjects
Brief Title: Safety, Pharmacokinetic, Pharmacodynamic Study of LAPS-IFNa in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11-HM10660A-101
Record Dates: First submitted 2011-12-27; First posted 2012-01-05 (Estimated); Last update posted 2014-02-07 (Estimated); Status verified 2014-02

CONDITIONS: Healthy
MeSH Terms: interventions — peginterferon alfa-2a

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- HM10660A (Experimental)
  Interventions: Biological: HM10660A
- Pegasys (Active Comparator)
  Interventions: Biological: Pegasys
- HM10660A Placebo (Placebo Comparator)
  Interventions: Biological: HM10660A placebo

INTERVENTIONS:
Biological: HM10660A — Single dose of HM10660A 1.5, 2.25, 3.0, or 4.0 ug/kg
  Arms: HM10660A
Biological: HM10660A placebo — Single dose of HM10660A Placebo
  Arms: HM10660A Placebo
Biological: Pegasys — Single dose of Pegasys 180ug
  Arms: Pegasys

SUMMARY:
Study design:

This is a randomized, double-blind, placebo- and active-controlled, single-dose study in 4 groups of 12 healthy male subjects each. In each group, 8 subjects will receive a dose of HM10660A, 2 subjects will receive a single dose of placebo and 2 subjects will receive a single dose of a currently marketed PEG-interferon.

DETAILED DESCRIPTION:
Primary objective:

to study the safety and tolerability of HM10660A, including immunogenicity, as compared to PEG-interferon alpha-2a

Secondary objective:

to study the pharmacokinetics and pharmacodynamics of HM10660A as compared to PEG-interferon alpha-2a

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 - 45 Years, Inclusive
* BMI: 18.0 - 28.0 kg/m2
* Are Non-smokers or Smoker of Fewer Than 5 Cigarettes Per Day as Determined by History

Exclusion Criteria:

* Mental Handicap
* Evidence of Clinically Relevant Pathology
* History of Type 1 Diabetes or Thyroid Disease

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2011-03; Primary Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Number of participants with AE occurrence, clinically significant clinical lab, vital sign, and/or ECG change | 43 days
  Number of participants with AE occurrence, clinically significant clinical lab, vital sign, and/or ECG change among HM10660A receivers will be assessed. It can be compared to those numbers in Active comparator group.

CONTACTS AND LOCATIONS:
Locations (1):
- Hanmi clinical, Netherlands, Netherlands